CLINICAL TRIAL: NCT04195256
Title: Intranasal Dexmedetomidine Plus Ketamine for Procedural Sedation in Children: an Adaptive Randomized Controlled Non-inferiority Multicenter Trial
Brief Title: Intranasal Dexmedetomidine Plus Ketamine for Procedural Sedation
Acronym: Ketodex
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Naveen Poonai (Other)
Responsible Party: Sponsor-Investigator, Naveen Poonai, Sponsor-Investigator/Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 091819
Record Dates: First submitted 2019-08-15; First posted 2019-12-11 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Fracture; Dislocation
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Adaptive, multi-centre, two-arm, randomized, blinded, double-dummy, controlled, parallel group, non-inferiority, phase II/III trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IN Ketodex (D4K2) (Experimental): Dexmedetomidine (Pfizer, Kirkland, Quebec), single-dose, 4 mcg/kg (0.04 mL/kg) of 100 mcg/mL solution, maximum of 200 mcg (2 mL) THEN Ketamine (Sandoz, Mississauga, Ontario), single dose, 2 mg/kg (0.04 mL/kg) of 50 mg/mL solution, maximum of 200 mg (4 mL) (D4K2), both delivered intranasally using a mucosal atomizer device (MAD) and divided to both nares AND 0.9% normal saline 0.03 mL/kg delivered intravenously to a maximum of 2 mL
  Interventions: Drug: IN Ketodex (D4K2)
- IN Ketodex (D3K3) (Experimental): Dexmedetomidine (Pfizer, Kirkland, Quebec), single-dose, 3 mcg/kg (0.03 mL/kg) of 100 mcg/mL solution, maximum of 200 mcg (2 mL) THEN Ketamine (Sandoz, Mississauga, Ontario), single dose, 3 mg/kg (0.06 mL/kg) of 50 mg/mL solution, maximum of 300 mg (6 mL) (D3K3), both delivered intranasally using a mucosal atomizer device (MAD) and divided to both nares AND 0.9% normal saline 0.03 mL/kg delivered intravenously to a maximum of 2 mL
  Interventions: Drug: IN Ketodex (D3K3)
- IN Ketodex (D2K4) (Experimental): Dexmedetomidine (Pfizer, Kirkland, Quebec), single-dose, 2 mcg/kg (0.02 mL/kg) of 100 mcg/mL solution, maximum of 200 mcg (2 mL) THEN Ketamine (Sandoz, Mississauga, Ontario), single dose, 4 mg/kg (0.08 mL/kg) of 50 mg/mL solution, maximum of 400 mg (8 mL) (D2K4), both delivered intranasally using a mucosal atomizer device (MAD) and divided to both nares AND 0.9% normal saline 0.03 mL/kg delivered intravenously to a maximum of 2 mL
  Interventions: Drug: IN Ketodex (D2K4)
- IV Ketamine (Active Comparator): Ketamine, single dose, 1.5 mg/kg (0.03 mL/kg) of 50 mg/mL solution delivered intravenously, to a maximum of 100 mg (2 mL) AND two aliquots of 0.9% normal saline in 3 possible combinations: (i) 0.04 mL/kg (max 2 mL) then 0.04 mL/kg (max 4 mL) (placebo D4K2), (ii) 0.03 mL/kg (max 2 mL) then 0.06 mL/kg (max 6 mL) (placebo D3K3), (iii) 0.02 mL/kg (max 2 mL) then 0.08 mL/kg (max 8 mL) (placebo D2K4), delivered intranasally using a MAD and divided to both nares
  Interventions: Drug: IV Ketamine

INTERVENTIONS:
Drug: IN Ketodex (D4K2) — Dexmedetomidine (Pfizer, Kirkland, Quebec), single-dose, 4 mcg/kg (0.04 mL/kg) of 100 mcg/mL solution, maximum of 200 mcg (2 mL) THEN Ketamine (Sandoz, Mississauga, Ontario), single dose, 2 mg/kg (0.04 mL/kg) of 50 mg/mL solution, maximum of 200 mg (4 mL) (D4K2), both delivered intranasally using a mucosal atomizer device (MAD) and divided to both nares AND 0.9% normal saline 0.03 mL/kg delivered intravenously to a maximum of 2 mL
  Other Names: Ketamine+Dexmedetomidine
  Arms: IN Ketodex (D4K2)
Drug: IN Ketodex (D3K3) — Dexmedetomidine (Pfizer, Kirkland, Quebec), single-dose, 3 mcg/kg (0.03 mL/kg) of 100 mcg/mL solution, maximum of 200 mcg (2 mL) THEN Ketamine (Sandoz, Mississauga, Ontario), single dose, 3 mg/kg (0.06 mL/kg) of 50 mg/mL solution, maximum of 300 mg (6 mL) (D3K3), both delivered intranasally using a mucosal atomizer device (MAD) and divided to both nares AND 0.9% normal saline 0.03 mL/kg delivered intravenously to a maximum of 2 mL
  Other Names: IN Ketodex II
  Arms: IN Ketodex (D3K3)
Drug: IN Ketodex (D2K4) — Dexmedetomidine (Pfizer, Kirkland, Quebec), single-dose, 2 mcg/kg (0.02 mL/kg) of 100 mcg/mL solution, maximum of 200 mcg (2 mL) THEN Ketamine (Sandoz, Mississauga, Ontario), single dose, 4 mg/kg (0.08 mL/kg) of 50 mg/mL solution, maximum of 400 mg (8 mL) (D2K4), both delivered intranasally using a mucosal atomizer device (MAD) and divided to both nares AND 0.9% normal saline 0.03 mL/kg delivered intravenously to a maximum of 2 mL
  Other Names: IN Ketodex III
  Arms: IN Ketodex (D2K4)
Drug: IV Ketamine — Ketamine, single dose, 1.5 mg/kg (0.03 mL/kg) of 50 mg/mL solution delivered intravenously, to a maximum of 100 mg (2 mL) AND two aliquots of 0.9% normal saline in 3 possible combinations: (i) 0.04 mL/kg (max 2 mL) then 0.04 mL/kg (max 4 mL) (placebo D4K2), (ii) 0.03 mL/kg (max 2 mL) then 0.06 mL/kg (max 6 mL) (placebo D3K3), (iii) 0.02 mL/kg (max 2 mL) then 0.08 mL/kg (max 8 mL) (placebo D2K4), delivered intranasally using a MAD and divided to both nares
  Other Names: Ketamine hydrochloride
  Arms: IV Ketamine

SUMMARY:
Orthopedic injuries comprise more than 10% of ED visits in children and 25 to 50% of children will sustain a fracture before age 16 years. Distal radius fractures account for 20-32% of fractures in children, making them the most common fracture type. Between 20 and 40% of extremity fractures in children require a closed reduction, often necessitating procedural sedation and analgesia (PSA). Intravenous (IV) ketamine is the most commonly used sedative agent used to perform a closed reduction. However, children rate IV insertion as the most painful hospital experience, second only to the injury itself. IV insertion can be more technically difficult in children because of smaller veins and lack of cooperation, often leading to multiple IV attempts. A combination of intranasal (IN) dexmedetomidine plus ketamine (IN Ketodex) may provide effective sedation for children undergoing a closed reduction without the distress and pain related to IV insertion. A less painful experience has been found to correlate with child satisfaction which may reduce caregiver anxiety and improve the therapeutic relationship with the health care team. This study is a multi-centre, two-arm, randomized, blinded, controlled, non-inferiority trial designed to test the hypothesis that IN Ketodex is non-inferior to intravenous (IV) ketamine with respect to depth of sedation as measured using the Pediatrics Sedation State Scale (PSSS).

DETAILED DESCRIPTION:
Intranasal medications may offer a technically easier and pain-free approach to procedural sedation (PSA); one that may have widespread applicability in patients with needle-phobia, difficult IV access, resource-limited settings, or when experience placing an IV is limited. Although IN ketamine has been found to be effective for fracture pain, procedural pain, anesthetic pre-induction, and diagnostic imaging, a recent shortage of this agent in the highest concentration of 100 mg/mL has severely limited out ability to study its effectiveness and consequent clinical uptake. Our research team conducted three systematic reviews of randomized trials of IN ketamine and IN dexmedetomidine in children undergoing painful procedures. The latter review included 18 trials (n=2128) of children age 1 month to 14 years. Our review found that IN dexmedetomidine, dosed from 1-4 mcg/kg, was well tolerated and superior to conventional sedatives (midazolam and chloral hydrate) in providing adequate sedation to 525/669 (78.5%) children. A number of studies found that IN dexmedetomidine was in fact superior to IN ketamine. Surendar et al. found that IN dexmedetomidine at 1.5 mcg/kg facilitated successful sedation in 18/21 (86%) of children undergoing dental procedures and was more effective than IN ketamine 5 mg/kg. Gyanesh et al. found that the proportion of children with satisfactory IV sedation was greater with IN dexmedetomidine 1 mcg/kg compared to IN ketamine 5 mg/kg [47/52 (90%) versus 43/52 (83%), respectively]. Mostafa et al. found that IN dexmedetomidine 1 mcg/kg was more effective at facilitating caregiver separation than IN ketamine 5 mg/kg or IN midazolam 0.2 mg/kg [30/32 (92%) versus 22/32 (69%) versus 28/32 (88%), respectively]. Moreover, a combination of dexmedetomidine and ketamine appeared to be superior than either agent alone. Qiao et al. found that IN dexmedetomidine 2 mcg/kg and oral ketamine 3 mg/kg in children undergoing IV insertion was superior to both IN dexmedetomidine 2.5 mcg/kg and oral ketamine 6 mg/kg alone (80.1% versus 47.6% versus 68.3%, respectively). Bhat et al. found that a combination of IN dexmedetomidine 1 mcg/kg and IN ketamine 2 mg/kg versus IN dexmedetomidine 1 mcg/kg alone facilitated greater acceptance of face mask (67% versus 52%, respectively) and greater tolerance of caregiver separation (93% versus 89%, respectively) (38). We also found evidence that higher doses of IN dexmedetomidine were more effective. More specifically, at the higher end of the dosing range (1-4 mcg/kg), IN dexmedetomidine 3 mcg/kg was superior to IN ketamine 7 mg/kg; providing adequate sedation to 25/29 (86.3%) versus 23/29 (79.4%) of children undergoing IV insertion, respectively. A dose-finding study of IN dexmedetomidine in children < 3 years who were post-operative from cardiac surgery and were undergoing transthoracic echocardiography found an optimal median effective dose of 3.3 mcg/kg (range 2.72-3.78 mcg/kg). Taken together, our review suggests that the most effective and tolerable intranasal agent for procedural sedation for fracture reduction is a combination of IN dexmedetomidine 4 mcg/kg and IN ketamine 2-3 mg/kg. There is ample and ongoing evidence of suboptimal management for procedural pain in children, a high frequency of orthopedic injuries requiring IV placement for PSA, and a lack of evidence to support the use of strategies that reduce the pain of IVs. However, there are no studies that have shown the effectiveness of IN ketamine for fracture reduction in children. In order to provide robust evidence supporting an alternate approach that precludes the need for an IV in children undergoing PSA, the investigators propose a study to answer the important research question: In children presenting to the ED with an orthopedic injury requiring PSA, does IN Ketodex provide as effective sedation as IV ketamine?

ELIGIBILITY:
INCLUSION CRITERIA

General Criteria

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Deemed by treating physician to require procedural sedation

Specific criteria

1. Children presenting to the paediatric EDs of participating sites age 2-17 years
2. Weighing up to and including 100 kg
3. One of the following injuries:

   * Closed forearm fracture
   * Metacarpal or phalangeal fracture
   * Dislocation of a shoulder or elbow
   * Type II supracondylar fracture
4. Expected to not require more than one dose of IV sedative medication if they were not in the trial (as determined by the procedure physician and not including cast or splint application).
5. Both nares are fully patent
6. Physician plans to sedate patient

EXCLUSION CRITERIA

1. Previous hypersensitivity reaction to ketamine or dexmedetomidine including rash, difficulty breathing, hypotension, apnea, or laryngospasm;
2. Suspected globe rupture;
3. Concomitant traumatic brain injury with intracranial hemorrhage;
4. Uncontrolled hypertension;
5. Nasal bone deformity or septal deviation;
6. Poor English or French fluency in the absence of native language interpreter;
7. American Society of Anesthesiologists (ASA) class 3 or greater;
8. Previous diagnosis of schizophrenia or active psychosis as per the treating physician
9. Neuro-cognitive impairment that precludes informed consent, assent, or ability to self-report pain and satisfaction;
10. More than one fracture or dislocation requiring reduction;
11. Hemodynamic compromise as per the treating physician;
12. Glasgow coma score < 15;
13. Previous sedation with ketamine or hematoma block within 24 hours;
14. Fracture is comminuted or associated with a dislocation;
15. Participant has undergone a hematoma block within 24 hours;
16. Obstructive sleep apnea
17. Previous enrollment in the trial;
18. Suspected pregnancy
19. Congenital heart disease or known cardiac dysrhythmia
20. Known or suspected hepatic impairment
21. Known renal insufficiency
22. Uncorrected mineralocorticoid deficiency

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adequate sedation | Through study completion in the ED (4 hours)
  Adequate is defined as fulfillment of all three of the following criteria:
  (i) A Pediatric Sedation State Scale (PSSS) score of 2 or 3 for the duration of the procedure (defined for closed reduction as the interval of time from the first application of traction or manipulation of the injured limb for the purpose of anatomical realignment to the last application of a realigning force). The PSSS is scored from 0 to 5 in discrete integer values every 15 seconds. A score of 4 or 5 indicates under-sedation and a score of 0 or 1 indicates over sedation.
  (ii) No additional medication is given during the procedure for the purpose of sedation.
  (iii) The patient did not actively resist, cry, or require physical restraint for completion of the closed reduction.

SECONDARY OUTCOMES:
Length of stay | Through study completion in the ED (4 hours)
  Defined as the time recorded in the medical record between triage and discharge.
Time to wakening | Through study completion in the ED (4 hours)
  This will be defined as the duration of time between the first pair of IN sprays and the first PSSS score of > 3 post-closed reduction.
Adverse effects | Through study completion in the ED and up to 72 hours post-discharge
  Adverse effects as defined by Health Canada reporting standards

OTHER OUTCOMES:
Length of stay due to procedural sedation | Through study completion in the ED (4 hours)
  Defined as the time interval from the first pair of IN sprays/IV dose to discharge, reflective of the time difference associated with different routes of administration.
Duration of procedure | Through study completion in the ED (4 hours)
  Defined as time of the first pair of IN sprays to the end of cast or splint application (closed reduction) in minutes
Caregiver, participant, bedside nurse or respiratory therapist, and physician satisfaction | Through study completion in the ED (4 hours)
  Satisfaction will be measured using a visual analog scale (VAS) when the participant is deemed ready for discharge. The following questions will be posed: How satisfied were you with your child's sedation? (Caregiver if at bedside), How happy were you with your sleep? (Participant), or How satisfied were you with the level of sedation in your patient? (Sedating physician & nurse/respiratory therapist as per who is at bedside).
Nasal irritation | Through study completion in the ED (4 hours)
  Discomfort associated with nasal sprays will be assessed by the research nurse using the Faces Pain Scale -Revised (FPS-R) when the participant is deemed ready for discharge. The FPS-R is a self-report measure scored as either 0,2,4,6,8,10, with increasing numbers indicating greater pain.
Volume of IN intervention received / Volume of IN intervention intended | Through study completion in the ED (4 hours)
  Volume of IN intervention received / Volume of IN intervention intended
Adjunctive IV therapy and medications | Through study completion in the ED (4 hours)
  The number of participants requiring an IV for therapy unrelated to sedation (eg. analgesics, antibiotics, antiemetics, fluids) will be recorded.
Pre-sedation Pain | Through study completion in the ED (4 hours)
  Will be recorded by the research nurse from the participant using the Faces Pain Scale - Revised (FPS-R) immediately prior to the first pair of intranasal sprays
Patient Preference | Through study completion in the ED (4 hours)
  The following question will be posed to the child: "If you were to be put to sleep again for an injury, what would you prefer, an intravenous needle or nasal sprays (choose one)?"
Exploratory subgroup analyses | Through study completion in the ED (4 hours)
  A planned subgroup analyses to determine whether the between group difference in adequacy of sedation is dependent on (i) pain score prior to sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, Principal Investigator — Western University
Locations (6):
- Canada (6):
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Winnipeg Children's Hospital, Winnipeg, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heath A, Rios JD, Pullenayegum E, Pechlivanoglou P, Offringa M, Yaskina M, Watts R, Rimmer S, Klassen TP, Coriolano K, Poonai N; PERC-KIDSCAN Ketodex Study Group. The intranasal dexmedetomidine plus ketamine for procedural sedation in children, adaptive randomized controlled non-inferiority multicenter trial (Ketodex): a statistical analysis plan. Trials. 2021 Jan 6;22(1):15. doi: 10.1186/s13063-020-04946-3. PMID 33407719